CLINICAL TRIAL: NCT06243497
Title: Comparison of Cytokines Profile in Aqueous Humor and Tear Before and After UCP Treatment
Status: Recruiting | Type: Observational
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022KYPJ255
Record Dates: First submitted 2023-09-26; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2023-05

CONDITIONS: Glaucoma; Ultrasound Cyclo Plasty; Aqueous Humor; Tear; Cytokines
MeSH Terms: conditions — Glaucoma; Lacerations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Matched eyes: Patients with glaucoma matched by sex and age.
- Treated eyes with UCP: The patients were definitely diagnosed as glaucoma, No age or gender limitation, IOP(intraocular pressure) ≥ 21mmHg under the maximum tolerated dose of antiglaucoma medication, or IOP < 21mmHg and glaucomatous optic nerve damage progressed. UCP treatment is required for the patients.
  Interventions: Procedure: Ultrasound CycloPlasty

INTERVENTIONS:
Procedure: Ultrasound CycloPlasty — All procedures were performed using the EyeOP1 device . The coupling cone was placed and adjusted on the centre of the patient's eye by visualising an equal white scleral ring surrounding the cornea. The coupling cone was kept in place via vacuum suction activated using a foot pedal and was then filled with a balanced salt solution to allow ultrasound transmission. The transducers were automatically activated at a frequency of 21 MHz and an acoustic power of 2.45 W, with an 8-s duration for each sector and a 20-s pause between each treatment to allow complete evacuation of heat.
  Groups: Treated eyes with UCP

SUMMARY:
Glaucoma is the leading cause of irreversible vision loss in people aged 50 years and older worldwide, second only to cataracts. Ultrasound Cyclo Plasty was first proposed as a new minimally invasive technique in the 1980 s. In recent years, many clinical studies at home and abroad have confirmed the effectiveness, safety and repeatability of UCP. The ciliary body is the target organ of UCP, and the range and accuracy of intraoperative destruction of the ciliary body are the key factors affecting the success or failure of the operation. The production of aqueous humor is closely related to the ciliary body. The dynamic balance of its production and discharge can affect IOP, and its content can directly reflect the intraocular environment. Besides,tears are easy to collect and can be used for follow-up. Previous studies have shown that various proteins in aqueous humor or tear can provide a basis for the pathophysiological changes of glaucoma, and can also be a potential biomarker for predicting the success of anti-glaucoma surgery.

At present, UCP related research focuses on its effectiveness and safety, mainly reflected in three aspects : postoperative intraocular pressure, number of anti-glaucoma drugs and complications, and lack of relevant indicators that directly reflect postoperative intraocular environment changes. The purpose of this study was to reveal the changes of cytokines in aqueous humor after UCP in patients with primary glaucoma, to analyze the possible causes of these factors, and to speculate the effect of their interaction on the surgical effect, in order to increase the predictability of UCP procedure.

ELIGIBILITY:
Inclusion Criteria:

* The patient was definitely diagnosed as glaucoma, No age or gender limitation, IOP(intraocular pressure) ≥ 21mmHg under the maximum tolerated dose of antiglaucoma medication, or IOP < 21mmHg and glaucomatous optic nerve damage progressed.

Exclusion Criteria:

* Other eye diseases that could affect IOP; preoperative use of systemic steroid drugs; history of other anti-glaucoma surgery within 3 months; ocular infection 2 weeks prior to UCP

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inpatient sample
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Cytokine profiles(pg/ml) | through study completion, an average of 2 year
  Cytokine antibody array was used to detect cytokines in AH samples from UCP treatment group and control group. The analysis method is based on the principle of double antibody sandwich immunoassay, and 60 ul of samples are applied on each block. Antibodies against the selected cytokines were immobilized at specific locations on the chip surface. The cytokines in the sample were captured by the corresponding antibody, and a mixture of biotinylated antibodies was added to detect the binding cytokines. Finally, the signal was visualized using a fluorescent dye ( cy3 equivalent ) that binds to streptavidin. The InnoScan 300 Microarray Scanner ( Innopsys, Parc d 'Activités Activestre, Carbonne, France ) was used for fluorescent dye detection.
Intraocular pressure(mmHg) | through study completion, an average of 2 year
  Using non-contact tonometer (NCT) to measure intraocular pressure
Anterior segment parameters(mm) | through study completion, an average of 2 year
  Measured by ultrasound biomicroscopy, parameters included WTW, ciliary body length, ciliary process length and density.

SECONDARY OUTCOMES:
LogMAR visual acuity | through study completion, an average of 2 year
  Using Snellen visual acuity chart to measure naked eye vision and best corrected vision
Complications(n,%) | through study completion, an average of 2 year
  Including conjunctival congestion, corneal edema, corneal epithelial defect, anterior chamber inflammation, pupil deformation,cataract development/progression, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Chengguo Zuo, M.D,Ph.D, Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No